CLINICAL TRIAL: NCT05624957
Title: Efficacy of Lidocaine Saline Irrigation in Patients Undergoing Shoulder Arthroscopy: Randomized Controlled Study
Brief Title: Lidocaine Irrigation in Shoulder Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Hassan Mokhtar Elshorbagy Hetta, lecturer of anesthesia and ICU, Minia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 475:10/2022
Record Dates: First submitted 2022-11-03; First posted 2022-11-22 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Postoperative Pain; Analgesia
Keywords: Postoperative pain; Lidocaine; Shoulder arthroscopy
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- lidocaine (Experimental): The patients will undergo shoulder arthroscopy with lidocaine epinephrine fluids irrigation.
  Interventions: Drug: Lidocaine epinephrine
- control group (Placebo Comparator): The patients will undergo shoulder arthroscopy with epinephrine fluids irrigation only.
  Interventions: Drug: Epinephrin

INTERVENTIONS:
Drug: Lidocaine epinephrine — Under aseptic condition every one litre of fluid irrigation will be mixture with 10 ml of lidocaine 2% and 0.25mg epinephrine and the last one use before end of surgery dexamethasone 8 mg will be added.
  Arms: lidocaine
Drug: Epinephrin — 0.25 mg epinephrine mixed with one litre of fluid irrigation
  Arms: control group

SUMMARY:
Arthroscopic shoulder surgery is often associated with severe postoperative pain that is often significant enough to interfere with initial recovery and rehabilitation. The pain that can be difficult to manage without large dose of opioid.

The study aim to explore the effect of continuous irrigation of fluids mixed with lidocaine and epinephrine for analgesic consumption and postoperative pain after shoulder arthroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-60
* Both genders
* Shoulder arthroscopy
* ASA I-III

Exclusion Criteria:

* Drug allergy
* Psychiatric disorder
* Opioid dependence
* Liver disease
* Patient refuse

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-11-25 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
total analgesic consumption | 24 hours
  total nalbuphine consumed one day after surgery

SECONDARY OUTCOMES:
first analgesic request | 24 hours
  time of PCA request
Visual analogue pain score | 24 hours
  pain intensity at rest and movement from 0-10 which 0 no pain and 10 the worst pain

CONTACTS AND LOCATIONS:
Overall Officials: hassan m. hetta, lecturer, Principal Investigator — Minia University, faculty of medicine
Locations (1):
- Minia University Hospital, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No